CLINICAL TRIAL: NCT02384096
Title: COVERAGE - A Study to Evaluate the Effect of Precision Spectra™ SCS System's Programming Features and Lead Options on Patient Outcomes
Brief Title: A Study to Evaluate the Effect of Precision Spectra™ Programming Features and Lead Options on Patient Outcomes
Acronym: COVERAGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 90968587
Record Dates: First submitted 2015-01-28; First posted 2015-03-10 (Estimated); Results first posted 2018-07-19 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain
Keywords: stimulation; implantable; pulse generator; back pain; chronic pain; leg pain
MeSH Terms: conditions — Chronic Pain; Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Programming, then Advanced Programming (Active Comparator): Precision Spectra SCS System with CoverEdge Surgical Lead or more than 2 percutaneous leads. Subjects first received conventional single source programming followed by Precision Spectra SCS System advanced programming.
  Interventions: Device: Conventional single source programming; Device: Precision Spectra SCS System advanced programming
- Advanced Programming, then Conventional Programming (Active Comparator): Precision Spectra SCS System with CoverEdge Surgical Lead or more than 2 percutaneous leads. Subjects first received Precision Spectra SCS System advanced programming followed by conventional single source programming.
  Interventions: Device: Conventional single source programming; Device: Precision Spectra SCS System advanced programming

INTERVENTIONS:
Device: Conventional single source programming — Precision Spectra SCS System using conventional single source programming.
Device: Precision Spectra SCS System advanced programming — Precision Spectra SCS System using advanced programming

SUMMARY:
The study is a prospective, on-label, multi-center, blinded, randomized controlled trial with a cross-over design to evaluate the effect of Precision Spectra™ SCS System's programming features and lead options.

DETAILED DESCRIPTION:
The study is a sub-study of RELIEF - A Global Registry to Evaluate Long-Term Effectiveness of Neurostimulation Therapy for Pain (NCT01719055). The treatment will consist of permanent implant of a Precision Spectra™ SCS IPG with either a 32 contact CoverEdge™ Surgical Lead or with more than 2 percutaneous leads after a successful trial. Programming features and lead options of the Precision Spectra™ SCS System will be evaluated up to 3 months post-IPG activation. Following completion of the 3 month visit, subjects will continue to be followed for up to 36 months per the study requirements of the RELIEF Registry.

ELIGIBILITY:
Inclusion Criteria:

* Meets RELIEF Registry criteria for inclusion
* Primary complaint of persistent or recurrent low back pain, with or without leg pain
* Signed a valid, IRB/EC-approved informed consent form

Exclusion Criteria:

* Meets any RELIEF Registry criteria for exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Lechleiter, M.S., Study Director — Boston Scientific Neuromodulation Corporation
Locations (4):
- United States (4):
  - Physicians Research Group, LLC, Phoenix, Arizona
  - Albany Medical Center, Albany, New York
  - PCPMG Clinical Research Unit, LLC, Greenville, South Carolina
  - Spine Team Texas, Rockwall, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 subjects were enrolled in the study. 5 were withdrawn prior to randomization: 4 were withdrawn as failing to meet inclusion criteria and 1 at the subject's request prior to randomization. 12 were randomized, but 1 was randomized in error and was withdrawn same day. Statistically relevant conclusions cannot be made from this small sample size.
Groups:
- Conventional Programming, Then Advanced Programming: Precision Spectra SCS System with CoverEdge Surgical Lead. Subjects were randomized to first receive conventional single source programming followed by Precision Spectra SCS System advanced programming.
  Conventional single source programming: Precision Spectra SCS System using conventional single source programming.
  Precision Spectra SCS System advanced programming: Precision Spectra SCS System using advanced programming.
- Advanced Programming, Then Conventional Programming: Precision Spectra SCS System with CoverEdge Surgical Lead. Subjects were randomized to first receive Precision Spectra SCS System advanced programming followed by conventional single source programming.
  Conventional single source programming: Precision Spectra SCS System using conventional single source programming.
  Precision Spectra SCS System advanced programming: Precision Spectra SCS System using advanced programming.
Period: First Intervention (7 Days)
Arm/Group | Conventional Programming, Then Advanced Programming | Advanced Programming, Then Conventional Programming
Started | 5 | 7
Completed | 4 | 7
Not Completed | 1 | 0
Period: Second Intervention (7 Days)
Arm/Group | Conventional Programming, Then Advanced Programming | Advanced Programming, Then Conventional Programming
Started | 4 | 7
Completed | 4 | 6
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Programming, Then Advanced Programming | Advanced Programming, Then Conventional Programming | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 1 | 6 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Paresthesia Coverage ≥50%
Description: Paresthesia Coverage assesses how much of the subject's painful areas are covered by SCS-induced paresthesia. The number of subjects reporting paresthesia coverage ≥50% is reported.
Time Frame: 7, 14 days post activation
Population: All subjects who completed the day 7 and day 14 post-activation study visits were included. Statistical analysis was not performed as the sample size is too small to draw any statistically relevant conclusions.
Measure: Number; unit: Participants
Arm/Group | Conventional Programming, Then Advanced Programming | Advanced Programming, Then Conventional Programming
Number analyzed (Participants) | 4 | 7
Participants
  Advanced Programming | 3 | 5
  Conventional Programming: number analyzed (Participants) | 4 | 6
  Conventional Programming | 3 | 5

ADVERSE EVENTS:
Time Frame: From informed consent through completion of study (approximately 3 months)
Description: Arms/groups are combined instead of reported per intervention because subjects received both programming types (arms) in this crossover study. Additionally, adverse events did not necessarily occur when a subject was receiving one of the two programming types.
Groups:
- All Enrolled Subjects: Rate of device-related adverse events (AEs) and Serious Adverse Events (SAEs) are reported for 17 enrolled subjects from informed consent through completion of study.
Arm/Group | All Enrolled Subjects
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 2/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=17)
Infection (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Mid back muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days